CLINICAL TRIAL: NCT04649840
Title: Estimation of Dynamics of Humoral and Cellular Immunity in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other); The Republican Research and Practical Center for Epidemiology and Microbiology (Other)
Responsible Party: Sponsor
Other Study IDs: IBCE_COVID19_Immunity
Record Dates: First submitted 2020-12-01; First posted 2020-12-02 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Covid19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Immunity, Cellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 moderate: moderate COVID-19 associated pneumonia
  Interventions: Diagnostic Test: Humoral and cellular immunity
- COVID-19 severe: severe COVID-19 associated pneumonia
  Interventions: Diagnostic Test: Humoral and cellular immunity

INTERVENTIONS:
Diagnostic Test: Humoral and cellular immunity — Humoral (IgG) and cellular (antigen-specific cells) immunity

SUMMARY:
The goal of the project: to study the dynamics of the humoral and cellular immunity in patients after pneumonia caused by the SARS-CoV-2 virus at different time intervals, in order to predict the duration of immune protection

DETAILED DESCRIPTION:
* to form study groups of patients (at least 60 patients in total) who have recovered from pneumonia of varying severity caused by the SARS-CoV-2 virus (at least 30 patients in each of the groups of patients who have had pneumonia in moderate and severe forms);
* to investigate the parameters of cellular immunity (the content of antigen-specific T-cells to the main viral antigens - proteins S, N, M) in patients of different groups included in the trials, in dynamics 3, 6, 9 and 12 months after the COVID-19-associated pneumonia;
* to investigate the indicators of humoral immunity (the content of IgG to the main viral antigens - proteins S, N, M) in patients of different groups included in the trials, in dynamics 3, 6, 9 and 12 months after the COVID-19-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* patients recovered from the COVID-19 associated pneumonia (moderate and severe) in 1-3 month interval before inclusion into the trial;

Exclusion Criteria:

* cancer;
* drug and alcohol addiction;
* autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recovered from the COVID-19 associated pneumonia (moderate and severe)
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
The dynamics of humoral and cellular immunity | 1 year
  The dynamics of both humoral and cellular immunity in response to COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, MD, PHD, Study Director — Director
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus